CLINICAL TRIAL: NCT04833192
Title: The Cross-sectional Study and Longitudinal Study of the Diagnostic Efficiency of Serum Dehydroepiandrosterone Sulfate in Subclinical Hypercortisolism
Brief Title: Evaluation of New Diagnostic Indicator of Subclinical Hypercortisolism
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Dalong Zhu, Chief Physician, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Other Study IDs: LP2021
Record Dates: First submitted 2021-01-24; First posted 2021-04-06 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Adrenal Incidentaloma; Subclinical Hypercortisolism
Keywords: serum dehydroepiandrosterone sulfate; adrenocorticotropic hormone; surgical management; conservative management
MeSH Terms: conditions — Adrenal incidentaloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year

GROUPS / COHORTS (2):
- experimental group: patients diagnosed with subclinical hypercortisolism as assessed by an endocrinologist.
  Interventions: Diagnostic Test: experimental group
- control grpup: patients diagnosed with nonfunctional adrenal adenoma as assessed by an endocrinologist.

INTERVENTIONS:
Diagnostic Test: experimental group — DHEAS.24h-UFC,ACTH and cortisol are measured in the experimental group
  Groups: experimental group

SUMMARY:
The purpose of this study is to evaluate the serum dehydroepiandrosterone sulfate in subclinical hypercortisolism

DETAILED DESCRIPTION:
In the past few years, with the widespread use of chest and abdominal imaging, the prevalence of adrenal incidentaloma (AIs) has been increasing and now approaches the 8.7% incidence reported in autopsy series. subclinical hypercortisolism (SH) is noted in up to 30% of patients with adrenal incidentalomas. Several groups have reported adverse clinical sequelae in individuals with SH, with recent studies highlighting an increase in cardiovascular morbidity and mortality compared to the general population. Accurate exclusion or confirmation of a diagnosis of SH is therefore a key step in the investigation and management of patients with AIs. Suppressed adrenocorticotropic hormone (ACTH) and low dehydroepiandrosterone sulfate (DHEAS) levels are frequently found in SH patients. Present study added new evidence for the limitations of ACTH and confirmed the usefulness of DHEAS for the detection of SH especially with unsuppressed ACTH in AI patients. On one hand, in the cross-sectional study, biometric measurements and sex hormones (including DHEAS, 24h-UFC, ACTH and cortisol) are analysed to explore the differences among SH patients, and nonfunctional adrenal adenoma patients. One the other hand, in the longitudinal study, changes in DHEAS, ACTH and cortisol in SH with surgical management and SH with conservative management both at baseline and different follow-up months after their different treatment management are collected to explore the changes of DHEAS and ACTH of SH patients.

ELIGIBILITY:
Inclusion Criteria:

* patients with adrenal accidental tumor (diameter > 1cm) found by physical examination or imaging examination due to non-adrenal diseases

Exclusion Criteria:

* concomitant use of drugs influencing glucocorticoid metabolism or secretion
* major psychiatric illness or history of excess alcohol intake
* overt clinical features of hypercortisolism
* clinical and endocrine function evaluation (surgery patients at the same time reference to postoperative pathology) revealed primary aldosteronism, pheochromocytoma, adrenocortical carcinoma, adrenal metastasis of cancer, myelolipoma; oncocytoma, congenital adrenal cortex hyperplasia and ganglion cells neuroma/paraganglioma, schwannoma, adrenal hematoma and uncertain diagnosis)
* non-adenoma lesions such as cysts and hemorrhage
* The pregnancy
* Patients with severe underlying diseases (such as liver and kidney failure, acute severe infection, etc.) that may affect the function of the hypothalamus-pituitary-adrenal axis (HPA axis)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: subclinical hypercortisolism and adrenal nonfunctional adenoma patients
Sampling Method: Probability Sample
Enrollment: 202 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
The gender and age of the participants | 1 day
  age in years and sex (female or male) of patients
Participant's weight and height | 1 day
  BMI(body mess index) in kg/m^2= (weight in kg) /(height in m)^2
the diurnal rhythm of ACTH | 2 day
  plasma ACTH in pmol/L at 8:00 am, 16:00 pm and 24:00 midnight
the the diurnal rhythm of cortisol | 2 day
  serum cortisol in nmol/L at 8:00 am, 16:00 pm and 24:00 midnight measured on the same day as plasma ACTH
Patients' baseline DHEAS level | 1 day
  serum DHEAS in ug/dL
CT imaging of adrenal tumor | 1 day
  diameter in cm of adrenal adenoma
dexamethasone suppression test | 2 day
  Dexamethasone 1mg (0.75mg/ tablet, 1.5 tablets) was taken orally at 24:00 midnight, and plasma ACTH in pmol/L and serum cortisol in cortisol levels were measured by blood sample at 8:00 the next day

SECONDARY OUTCOMES:
the changes of DHEAS after surgical management | 1,3,6 and12 months after the surgical management (for subclinical hypercortisolism with surgical managment)
  DHEAS in ug/dL
the changes of ACTH after surgical management | 1,3,6 and12 months after the surgical management (for subclinical hypercortisolism with surgical managment)
  ACTH in pmol/L
the changes of cortisol after surgical management | 1,3,6 and12 months after the surgical management (for subclinical hypercortisolism with surgical managment)
  cortisol in nmol/L
the changes of DHEAS after conservative management | 12 months after the conservative management (for subclinical hypercortisolism with conservative management)
  DHEAS in ug/dL
the changes of ACTH after conservative management | 12 months after the conservative management (for subclinical hypercortisolism with conservative management)
  ACTH in pmol/L
the changes of cortisol after conservative management | 12 months after the conservative management (for subclinical hypercortisolism with conservative management)
  cortisol in nmol/L

CONTACTS AND LOCATIONS:
Locations (1):
- at Divison of Endocrinology,the Affiliated Drum Tower Hospital of Nanjing University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu MS, Lou Y, Chen H, Wang YJ, Zhang ZW, Li P, Zhu DL. Performance of DHEAS as a Screening Test for Autonomous Cortisol Secretion in Adrenal Incidentalomas: A Prospective Study. J Clin Endocrinol Metab. 2022 Apr 19;107(5):e1789-e1796. doi: 10.1210/clinem/dgac072. PMID 35137142